CLINICAL TRIAL: NCT05785143
Title: Utilizing Dry Lab Database to Analyze the Prognostic Factors of Multi-trauma Patients and Determine the Optimal Timing of Definitive Orthopedic Operation
Brief Title: Timing of Damage Control Orthopedic Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH111-REC2-110
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: The Precision Personal Timeline in Definitive Surgery Associated With Outcome
Keywords: multi-trauma; lactate; definitive orthopedic operation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Utilizing dry lab database to analyze the prognostic factors of multi-trauma patients and determine the optimal timing of definitive orthopedic operation — to analyze if serum lactate a predictive factor of optimal surgical timing in multi-trauma patients. In order to obtain more accurate data, we choose to utilize ili database and trauma database instead of National Health Insurance Research Database.

SUMMARY:
The decision to operate and surgical timing on multi-trauma patients remains controversial, inappropriate surgical timing may cause more complications which lead to poor prognosis. We hope to find out the connection between lactate and prognosis in multi-trauma patients, and the optimal timing of definitive treatment.

DETAILED DESCRIPTION:
The decision to operate and surgical timing on multi-trauma patients remains controversial, inappropriate surgical timing may cause more complications which lead to poor prognosis.

The aim of our study is to analyze if serum lactate a predictive factor of optimal surgical timing in multi-trauma patients. In order to obtain more accurate data, we choose to utilize ili database and trauma database instead of National Health Insurance Research Database.

Multi-trauma patients from 2002 through 2022 were included to our study. We hope to find out the connection between lactate and prognosis in multi-trauma patients, and the optimal timing of definitive treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) Injury severity score(ISS) > 16 with pelvicfracture or long bone fracture requiring surgical fixation (2) Patient age ≥ 20. Pathologic fracture was excluded. Our primary endpoint si mortality rate, secondary endpoints include ICU stay, ICU complications (Sepsis, Pneumonia, Multiple organ failure)

Exclusion Criteria:

* death before into undergoing surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pelvic fracture patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
EQ5D5L | 1 year
  The functional outcome of daily activity

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan